CLINICAL TRIAL: NCT07199322
Title: Clinical validatiOn of an AI-based DEcision Support System for Robotic Upper Limb Rehabilitation in Patients With Stroke. A CO-AIDER Study.
Acronym: COAIDER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Policlinico Universitario Campus Bio-Medico (Other); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COAIDER; RF-2021-12375472 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Stroke Ischemic; Stroke Hemorrhagic; Upper Limb Rehabilitation
Keywords: Stroke; Upper limb rehabilitation; Artificial Intelligence; Robot-assisted therapy; AI-supported robotic system; AI-based decision support system; rehabilitation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, controlled, two-arm clinical study of a non-CE-marked medical device for non-commercial purposes. Participants will be randomly assigned to either robotic rehabilitation supported by the AI-DSS (software CO-AIDER) or robotic rehabilitation with treatment parameters set by clinical staff.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic treatment with an AI-based decision support system (Robotic therapy + CO-AIDER software) (Experimental): Participants assigned to this arm will receive upper limb robotic treatment using the MOTORE robotic device, supported by the AI-based decision support system (CO-AIDER software). CO-AIDER implements a predictive model based on recurrent neural networks (LSTM) that analyzes demographic, clinical, and kinematic data collected during treatment sessions. The model estimates the expected post-treatment scores on three standard clinical scales (FMA, ARAT, and MI). In addition to outcome prediction, the system provides therapists with recommendations on robot parameters (stiffness, weight, and viscosity), which are used to personalize the difficulty level of the exercises implemented in MOTORE, without directly altering the therapeutic course.
  Interventions: Device: Robotic upper limb rehabilitation in patients with Stroke with AI support
- Robotic treatment with parameters defined exclusively by the clinical team (Robotic Therapy) (Active Comparator): Participants assigned to the control group will receive upper limb robotic treatment using the MOTORE robotic device. The treatment will be identical to the experimental arm in terms of device and exercise types, but all parameters will be determined exclusively by the physiotherapists based on their clinical expertise, without AI-based decision support.
  Interventions: Device: Robotic upper limb rehabilitation in patients with Stroke without AI support

INTERVENTIONS:
Device: Robotic upper limb rehabilitation in patients with Stroke with AI support — Participants will receive upper limb robotic treatment using MOTORE (Mobile robot for upper limb neurOrtho Rehabilitation), a medical device indicated for post-stroke and post-traumatic rehabilitation. MOTORE is a portable, autonomous, omnidirectional, haptic robot that provides force feedback to the user and supports active, passive, and assistive movements.
  The device includes software with assessment and rehabilitation exercises presented as interactive games (serious games), enabling personalized therapy and measurement of patient performance. MOTORE follows the "assist as needed" paradigm, actively assisting or resisting movements based on the patient's intentions. Parameters are set by the AI-based decision support system (CO-AIDER). Treatment will be delivered daily for 45 minutes, five days per week, for a total of 30 sessions.
  Other Names: RT + COAIDER; Robotic Therapy + COAIDER
  Arms: Robotic treatment with an AI-based decision support system (Robotic therapy + CO-AIDER software)
Device: Robotic upper limb rehabilitation in patients with Stroke without AI support — Participants will receive upper limb robotic treatment using MOTORE (Mobile robot for upper limb neurOrtho Rehabilitation), a medical device indicated for post-stroke and post-traumatic rehabilitation. MOTORE is a portable, autonomous, omnidirectional, haptic robot that provides force feedback to the user and supports active, passive, and assistive movements.
  The device includes software with assessment and rehabilitation exercises presented as interactive games (serious games), enabling personalized therapy and measurement of patient performance. MOTORE follows the "assist as needed" paradigm, actively assisting or resisting movements based on the patient's intentions. Parameters are set by the clinical team based on their expertise. Treatment will be delivered daily for 45 minutes, five days per week, for a total of 30 sessions.
  Other Names: Robotic Therapy; RT
  Arms: Robotic treatment with parameters defined exclusively by the clinical team (Robotic Therapy)

SUMMARY:
The goal of this clinical trial is to validate an artificial intelligence-based decision support system (AI-DSS) for robotic rehabilitation in participants with stroke.

The study aims to answer the following questions:

* Can the AI-DSS support therapists in setting therapy parameters and adapting personalized robotic rehabilitation programs effectively?
* Can AI-supported robotic rehabilitation improve upper limb function, activities of daily living (ADL), cognitive function, and quality of life compared with standard therapist-guided robotic rehabilitation?

Researchers will compare two groups:

* Robotic rehabilitation supported by the AI-DSS (CO-AIDER);
* Robotic rehabilitation with parameters set by therapists (control group).

Participants will:

* Receive robotic rehabilitation for the upper limb, either guided by the AI-DSS or by therapists;
* Be monitored throughout the program, with therapy parameters adjusted according to their progress;
* Complete assessments to evaluate changes in upper limb function, activities of daily living, cognitive function, and quality of life.

The study will also evaluate the usability and acceptability of the AI-supported robotic system as perceived by participants and clinical staff, and will include a cost-effectiveness analysis of the two interventions.

DETAILED DESCRIPTION:
The CO-AIDER study is a multicenter, randomized, controlled, two-arm, non-profit clinical trial validating an AI-based decision support system (AI-DSS) in robotic upper limb rehabilitation for stroke patients. It supports therapists in setting therapy parameters and personalizing rehabilitation programs while monitoring patient progress. A total of 100 participants with ischemic or hemorrhagic stroke in the subacute phase (within six months of the event) will be randomly assigned to two groups. The experimental group will receive upper limb robotic rehabilitation using the MOTORE device supported by the AI-DSS CO-AIDER, which predicts motor recovery and provides recommendations for optimal therapy parameters based on clinical and instrumental data. Recommendations focus on stiffness, weight, and viscosity, key parameters for tailoring therapy to patients' abilities. The system provides guidance only and does not directly affect therapy progression. The control group will receive the same robotic treatment, with parameters set by therapists based on their clinical expertise. All participants will complete 30 sessions of robotic rehabilitation, 45 minutes per day, five days per week, alongside a conventional rehabilitation program for lower limbs and trunk. Assessments will be performed at baseline (T0, within 7 days of enrollment), mid-treatment (T1, after 15 sessions), and at the end of treatment (T2, after 30 sessions). Clinical assessment will include measures of upper limb motor function, activities of daily living, pain, spasticity, cognitive function, and quality of life using standardized clinical scales. Robotic performance will be assessed using parameters collected by the MOTORE system. Usability and acceptability of the AI-DSS will be evaluated through validated questionnaires. Randomization will be stratified by disease onset, motor impairment, and recruitment center to ensure balanced allocation. Data will be collected and stored pseudonymously in a secure, encrypted database. A cost-effectiveness analysis will compare AI-DSS-supported rehabilitation with therapist-guided therapy. The study will also evaluate how patients and clinical staff perceive the AI-supported robotic system in routine rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic stroke confirmed by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI);
* Age between 18 and 85 years;
* Time since stroke less than six months;
* Mild to severe upper limb impairment (Fugl-Meyer Assessment for Upper Extremity (FMA-UE) ≤ 58).

Exclusion Criteria:

* Behavioral or cognitive disorders and/or reduced compliance;
* Severe spasticity or hypertonia in the affected limb (Modified Ashworth Scale (MAS) > 3);
* Severe visual impairments;
* Concurrent participation in another clinical trial for upper limb rehabilitation following stroke;
* Refusal to provide written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Usability and acceptability for therapists | Baseline; during the study; within 48 hours from the end of the treatment
  Evaluation of usability and acceptability for therapists will be conducted through ad hoc questionnaires and the System Usability Scale (SUS). The SUS is a standardized tool developed to assess the perceived usability of systems, devices, or services. It consists of 10 items rated on a 5-point Likert scale, covering aspects such as ease of use, complexity, and learnability. The SUS provides a global usability score ranging from 0 to 100, where higher scores indicate better usability.
Change from baseline in the Fugl-Meyer Assessment for the upper extremities - motor function (FMA-UE) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The upper extremity motor function domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, and hand. It ranges from 0 (hemiplegia) to 66 (normal motor performance).

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The National Institutes of Health Stroke Scale (NIHSS) is a validated tool for assessing stroke severity. The score ranges from 0 to 42, with higher scores indicating more severe neurological deficit.
Motricity Index (MI) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Motricity Index (MI) is an ordinal method of measuring limb strength. For the upper extremity, shoulder abduction, elbow flexion, and pinch grip are considered; for the lower extremity, hip flexion, knee extension, and ankle dorsiflexion are considered. It ranges from 0 (worse) to 100 (normal strength).
Modified Ashworth Scale (MAS) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Modified Ashworth Scale (MAS) is a revised version of the original Ashworth Scale that measures spasticity in patients with lesions to the central nervous system. MAS is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0 to 4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch. The lower the score, the lower the spasticity. Upper and lower joints spasticity is assessed.
Douleur Neuropathique 4 (DN4) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Douleur Neuropathique 4 (DN4) questionnaire is a validated clinician-administered screening tool for neuropathic pain. It ranges from 0 to 10; higher values means higher neuropathic pain probability.
Numerical Rating Scale for Pain (NRS) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Numerical Rating Scale for Pain(NRS) is a tool used to assess pain intensity. It is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Modified Barthel Index (mBI) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The modified Barthel Index for Activities of Daily Living is a validated ordinal scale which measures a person's ability to complete activities of daily living (ADL). Scores range from 0 (total dependence) to 100 (total independence).
Frenchay Arm Test (FAT) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Frenchay Arm Test (FAT) assesses motor skills during activities of daily living (ADL) in patients with upper extremity impairments due to neurological conditions, using five practical tasks. Each task is scored 0 (unable) or 1 (able), for a total score of 0-5. Higher scores indicate better arm and hand function.
Action Research Arm Test (ARAT) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Action Research Arm Test (ARAT) is a 19 item observational measure used to assess upper extremity performance (coordination, dexterity and functioning). The 19 items comprising the ARAT are scored using a 4 point ordinal scale. Scores on the ARAT may range from 0-57 points, with a maximum score of 57 points indicating better performance.
Short-Form Health Survey (SF-36) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Short-Form Health Survey (SF-36) is a questionnaire that assesses a person's health status. It includes 36 items across eight domains: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional health, and mental health. Each domain is scored from 0 to 100, with higher scores indicating better health or functioning.
Montreal Cognitive Assessment (MoCA) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. It ranges from 0 (worst) to 30 (best).
Symbol Digit Modalities Test (SDMT) | Baseline (within 7 days of enrollment); within 48 hours from the 15th session; within 48 hours from the 30th session
  The Symbol Digit Modalities Test evaluates information processing speed. It consists of a simple task of replacing symbols with numbers. Using a reference key, the patient has 90 seconds to match a sequence of symbols with the correspondent numbers as rapidly as possible. Both written or oral administration can be used. For each correct answer, a point is assigned. The higher the score, the faster the information processing speed.
Cost-effectiveness analysis of CO-AIDER software | Baseline; within 48 hours from the 15th session; within 48 hours from the 30th session
  A cost-effectiveness analysis of the CO-AIDER software will be carried out in terms of the added value of the solution, defined as the ratio between Delta_Outcome (i.e., the difference in clinical outcomes obtained with and without the support of the CO-AIDER software) and Delta_Cost (i.e., the difference in treatment costs with and without the support of the CO-AIDER software).
Therapist satisfaction (Technology Acceptance Model, TAM) | Within 48 hours from the 30th session
  Assessment of therapist satisfaction and technology acceptance using the Technology Acceptance Model (TAM). The TAM is a questionnaire used with the primary aim of identifying the determinants involved in the acceptance of Robotic and Allied Technology. The questionnaire consists of 4 sections (perceived usefulness, ease of use, compatibility, intention to use); each question includes a 7-point Likert scale, from 1 (worst) to 7 (best). The scoring is calculated for each section and is given by the average of the responses in that section, ranging from 1 (worst) to 7 (best).
Patient satisfaction (Technology Acceptance Model, TAM) | Within 48 hours from the 30th session
  Assessment of patient satisfaction and technology acceptance using the Technology Acceptance Model (TAM). The TAM is a questionnaire used with the primary aim of identifying the determinants involved in the acceptance of Robotic and Allied Technology. The questionnaire consists of 4 sections (perceived usefulness, ease of use, compatibility, intention to use); each question includes a 7-point Likert scale, from 1 (worst) to 7 (best). The scoring is calculated for each section and is given by the average of the responses in that section, ranging from 1 (worst) to 7 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Guglielmelli, PhD, Study Chair — Campus Bio-Medico University; Irene G Aprile, MD, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi ONLUS, Roma
Locations (10):
- Italy (10):
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Sant'Angelo dei Lombardi, AV
  - Fondazione Don Carlo Gnocchi, Centro Spalenza, Rovato, BS
  - IRCSS Fondazione Don Carlo Gnocchi, Florence, FI
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Tricarico, Mount
  - Scuola Superiore Sant'Anna, Pisa, PI
  - Fondazione Don Carlo Gnocchi, Centro Gala, Acerenza, PZ
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma, RM
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria della Provvidenza, Roma, RM
  - Fondazione Don Carlo Gnocchi, Santa Maria dei Poveri Polo Riabilitativo del Levante ligure, La Spezia, SP
  - Fondazione Don Carlo Gnocchi, Centro Santa Maria ai Colli - Presidio Sanitario Ausiliatrice, Torino, TO

REFERENCES:
- [Background] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2018 Sep 3;9(9):CD006876. doi: 10.1002/14651858.CD006876.pub5. PMID 30175845
- [Background] Germanotta M, Cruciani A, Pecchioli C, Loreti S, Spedicato A, Meotti M, Mosca R, Speranza G, Cecchi F, Giannarelli G, Padua L, Aprile I. Reliability, validity and discriminant ability of the instrumental indices provided by a novel planar robotic device for upper limb rehabilitation. J Neuroeng Rehabil. 2018 May 16;15(1):39. doi: 10.1186/s12984-018-0385-8. PMID 29769127
- [Background] Aprile I, Germanotta M, Cruciani A, Loreti S, Pecchioli C, Cecchi F, Montesano A, Galeri S, Diverio M, Falsini C, Speranza G, Langone E, Papadopoulou D, Padua L, Carrozza MC; FDG Robotic Rehabilitation Group. Upper Limb Robotic Rehabilitation After Stroke: A Multicenter, Randomized Clinical Trial. J Neurol Phys Ther. 2020 Jan;44(1):3-14. doi: 10.1097/NPT.0000000000000295. PMID 31834217